CLINICAL TRIAL: NCT06569303
Title: Virtual Positive Parenting Intervention to Promote Filipino Family Wellness: A Randomized Controlled Trial : Filipino Family Health Initiative 1.0
Brief Title: Filipino Family Health Initiative 1.0
Acronym: FFHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of Southern California (Other); University of California, San Diego (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Joyce Javier, Associate Professor, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KPSOM-2189823; 7R01MD017003 (NIH); NCT06416423 (obsolete NCT alias)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety; Parenting
Keywords: Filipino Families; Incredible Years; Mental Health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents assigned to the intervention arm will receive the Incredible Years® School Age Basic & Advanced Parent Training Program. It consists of twelve (12) 2-hour online workshops led by a certified peer coach in the Incredible Years Parent Training Series.
  Interventions: Behavioral: Incredible Years® School Age Basic Parent Training Program
- Control (Other): Parents assigned to the control arm will be emailed and mailed written parent education materials from the American Academy of Pediatrics called the Bright Futures handouts. The control group is offered the Incredible Years® School Age Basic & Advanced Parent Training Program after a 3-month wait list period.
  Interventions: Behavioral: Incredible Years® School Age Basic Parent Training Program; Behavioral: American Academy of Pediatrics, Bright Futures Handouts

INTERVENTIONS:
Behavioral: Incredible Years® School Age Basic Parent Training Program — The Incredible Years® School Age Basic Parent Training Program targets many of the proposed mechanisms and risk factors for internalizing distress in early childhood: harsh and unpredictable or critical parenting behaviors. Parents also learn cognitive strategies; such as self-praise, coping thoughts, how to challenge negative thoughts, and how to get support that they are encouraged to model for and teach their children. Finally, the participants learn how to be more positive and nurturing through academic, social and emotional coaching.
Behavioral: American Academy of Pediatrics, Bright Futures Handouts — Written materials that include age-group specific tips on how parents can support their child's development and social and academic success.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an online parenting program on Filipino parents living in California. The main aims are to:

* Test the effectiveness of the online Incredible Years® model of parent training and its impact on primary outcomes.
* Determine the impact of intervention engagement (i.e., higher attendance) on parenting practices and child behavior outcomes.
* Describe Intervention delivery and its online implementation in real-world community settings.

The study involves two phases:

* Phase 1: Participants will receive the Online Incredible Years® School Age Basic & Advanced Parent Training Program (intervention) and complete parent-reported and child-reported measures at baseline, 3 months and 6 months.
* Phase 2: Parenting Group Leaders will each participate in one semi-structured interview to inform the sustainability of the intervention in real world community settings. Researchers will compare 250 Filipino families, half of which will receive the intervention and the other half will receive the American Academy of Pediatrics' Bright Futures handouts (control) and be placed on a 3-month waitlist for the IY parenting program. Both groups will be followed for a minimum of 6 months with follow- up assessments that include parent-report and child report measures.

DETAILED DESCRIPTION:
Evidence-based parenting interventions provided in early childhood have proven to be effective in preventing the onset and escalation of child mental health disorders. The overall objective of the proposed research is to test the effectiveness of a parenting program (Incredible Years® School Age Advance and Basic Parent Training Program, IYP) in Filipino parents recruited from multiple community-based settings and its impact on trajectories of parenting practices, parenting stress, and child problem behavior. IYP is one of the best studied and most highly regarded parent training programs.

Through pilot studies funded by an National Institutes of Health (NIH) Mentored Patient-Oriented Research Career Development Award (K23) and an National Center for Advancing Translational Sciences (NCATS) Mentored Career Development Award (KL2) award, the investigators identified IYP as a community-identified solution for preventing behavioral health problems, demonstrated IYP efficacy in improving parenting practices and parenting stress in Filipino parents, and child problem behavior. This population was chosen because: 1) Filipinos are the third largest Asian population in the U.S. with the highest concentration living in Los Angeles; 2) Filipinos are exposed to multiple adversities, including immigration stress and relocation, loss of social status, and lower self-esteem, placing young children at risk for future behavioral and mental health problems; 3) U.S.-born Filipino youth exhibit higher rates of mental health problems than non-Hispanic whites and attain significantly lower levels of education than their foreign-born counterparts and other U.S.-born Asian American populations; and 4) Filipinos are less likely than non-Hispanic whites to participate in mental health and preventive care interventions.

The sample will include 500 individuals, 250 Filipino parent-child dyads. Data will be obtained using process evaluation tracking system and self-report instruments. The specific aim is to test the effectiveness of the Incredible Years model of parent training and its impact on parenting practices (primary outcome). It is hypothesized that 1) Parents will report and demonstrate improvements in parenting practices after IYP, as compared to baseline and to the control condition; 2) Parents in the experimental group will show more rapid improvement in parenting practices and these effects will be sustained over time compared to those in the control condition; and 3) Parents will report improvements in parenting stress, child problem behavior, such as internalizing, externalizing, and depressive symptoms (secondary outcomes) after IYP as compared to baseline and to the control condition.

Findings will contribute to the scientific literature on preventive and early intervention programs for children at high risk for future behavioral problems. The data will also provide important information to understand the processes underlying how IYP affects parenting practices and subsequent child problem behavior among Filipino families. The importance of this research rests on its potential to prevent behavioral health disparities in this understudied and high-risk population.

The investigators also aim to describe intervention delivery and its online implementation in real-world community settings. Research Question 1: What are the facilitators/barriers to implementing the intervention at multiple levels (consumer, staff/provider, community setting)? Research Question 2: What are the facilitators and barriers to sustaining the intervention during and after the study?

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of at least one child 8-12 years of age
* Parent or legal guardian is of Filipino descent
* Parent or legal guardian and child are English speaking
* Pregnant women or legal guardians may be included if they have a child who meets the inclusion and exclusion criteria

Exclusion Criteria:

* Family plans to move out of the state of California within the next 6 months
* Family has previously participated in the Incredible Years (IY) curriculum
* Parent or legal guardian are not fluent in English
* Adults unable to consent or children unable to assent
* Prisoners

Note: All parent participants in the study are 18 years or older. Youth participants are 8-12 years old.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Parent Reported Positive Verbal Discipline | Baseline, 3 months, 6 months
  Parenting practices will be assessed using scores from the Parent Practices Interview (PPI). The PPI asks questions regarding parenting styles and behavior management techniques. Questions are rated on a scale ranging from never to always
Child Reported Depression Symptoms | Baseline, 3 months, 6 months
  Child depression will be measured using the Child Depression Inventory (CDI). Each item in this self-report instrument includes a list of sentences that describe how children typically feel. Children are asked to pick out the sentence that best describes how they feel over the past 2 weeks.
Child Reported Anxiety Symptoms | Baseline, 3 months, 6 months
  Child anxiety will be measured using the Screen for Child Anxiety Related Emotional Disorders (SCARED). Screen includes a list of sentences that describe how people feel over the last 3 months. Answers are rated on a scale from 0 (not true) to 2 (very true or often true).

SECONDARY OUTCOMES:
Parent Reported Use of Physical Punishment | Baseline, 3 months, 6 months
  Parent reported use of physical punishment will be assessed using scores from the Parent Practices Interview (PPI).
  The PPI asks questions regarding parenting styles and behavior management techniques. Questions are rated on a scale ranging from never to always.
Parent Reported Change in Child Behavioral Problems | Baseline, 3 months, 6 months
  Child problem behavior will be measured using scores from Child Behavior Checklist (CBCL). Parents describe their child's behavior within the past 6 months. Questions are rated on a scale from 0 (not true) to 2 (very true or often true). The CBCL screens for the following behaviors: Aggressive Behavior, Anxious/Depressed, Attention Problems, Rule-Breaking Behavior, Somatic Complaints, Social Problems, Thought Problems, Withdrawn/Depressed. Results for each subscale are presented as a percentile and T-score, with scores above 97th percentile considered as "clinical range" based on the Diagnostic and Statistical Manual of Mental Disorders (DSM)-V.
Parent Reported Child Anxiety | Baseline, 3 months, 6 months
  Parent reported child anxiety will be measured using scores from the Screen for Child Anxiety Related Disorders (SCARED). Screen includes a list of sentences that describe how people feel over the last 3 months. Answers are rated on a scale from 0 (not true) to 2 (very true or often true).
Parent Reported Child Depression | Baseline, 3 months, 6 months
  Parent Reported Child Depression will be measured using scores from the Children's Depression Inventory (CDI).
  Screen includes statements that describes observations of subject's child over the past 2 weeks. Answers are rated on a scale from 0 (not at all) to 3 (much or most of the time).
Parent Reported Child Resilience | Baseline, 3 months, 6 months
  Parent Reported Child Resilience will be measured using scores from the Child & Youth Resilience Measure- Revised Person Most Knowledgeable Version (PMK-CYRM-R). Questions include statements designed to better understand how the subject's child copes with daily life. Answers are rated on a scale from 1( not at all) to 5 (a lot).
Child Reported Child Resilience | Baseline, 3 months, 6 months
  Child Reported Child Resilience will be measured using scores from the Child & Youth Resilience Measure (CYRM-R).
  Questions include statements designed to better understand how the child copes with daily life. Answers are rated on a scale from 1( not at all) to 5 (a lot).
Parenting Self Efficacy | Baseline, 3 months, 6 months
  Parenting Self Efficacy will be measured using scores from the Parenting Sense of Competence (PSOC). Questions include agree/ disagree statements about perceived self efficacy and satisfaction with parenting. Answers are rated on a scale from 1( Strongly Disagree) to 6 (Strong Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Javier, MD MPH MS, Principal Investigator — Kaiser Permanente School of Medicine
Locations (1):
- Kaiser Permanente Bernard J. Tyson School of Medicine, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be provided to the NIH National Institute of Mental Health Data Archives (NDA) repository.
  The de-identified individual data will be shared with the NIH National Institute of Mental Health Data Archives (NDA) repository. Any information that could be used to identify you will be removed before any data is shared. NDA provides infrastructure for sharing research data, tools, methods, and analyses enabling collaborative science and discovery. De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.
  The NDA makes available human subjects data collected from hundreds of research projects across many scientific domains. De-identified human subjects data, harmonized to a common standard, are available to qualified researchers.
Time Frame: Data will be shared with authorized users upon publication (via an NDA Study) or 1-2 years after the grant end date specified on the first Notice of Award, as defined in the applicable Data Sharing Terms and Conditions.
  Specific data used in a publication will be shared at the time of publication. All other data that are part of the principal investigator's final dataset as defined in the Data Sharing Terms and Conditions will be shared 2 years after the original project end date.
Access Criteria: Researchers studying parenting and child behavior outcomes.
URL: https://nda.nih.gov/

REFERENCES:
- [Result] Javier JR, Aguiling W, Cunanan P, Sepulveda A, Coffey DM, Castro J, Palinkas LA, Kipke MD, Mack WJ. Short-term outcomes from a pilot randomized controlled trial evaluating a virtual culturally adapted parenting intervention among Filipino parents of school-age children. Cultur Divers Ethnic Minor Psychol. 2025 Jan;31(1):124-137. doi: 10.1037/cdp0000616. Epub 2023 Oct 19. PMID 37856386